CLINICAL TRIAL: NCT00069082
Title: A Phase III, Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Multicenter Evaluation of Civamide (Zucapsaicin) Nasal Solution in the Treatment of Episodic Cluster Headache
Brief Title: Intranasal Civamide for Episodic Cluster Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Winston Laboratories (Industry)
Responsible Party: Scott B. Phillips, M.D., Study Director, Winston Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WL-1001-02-05
Record Dates: First submitted 2003-09-15; First posted 2003-09-16 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Episodic Cluster Headache
Keywords: Headache; Cluster; EC; Episodic Cluster
MeSH Terms: conditions — Cluster Headache; Headache | interventions — zucapsaicin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Civamide (Active Comparator): Nasal Solution 0.01%
  Interventions: Drug: Civamide (Zucapsaicin)
- Placebo (Placebo Comparator): Placebo nasal solution with sodium chloride 10%
  Interventions: Drug: Sodium Chloride

INTERVENTIONS:
Drug: Civamide (Zucapsaicin) — Nasal Solution 0.01%
  Arms: Civamide
Drug: Sodium Chloride — Nasal Solution 10%
  Arms: Placebo

SUMMARY:
This is a 49-day study to evaluate the effectiveness of Intranasal Civamide (Zucapsaicin) in the treatment of an episodic cluster headache period compared to placebo (medically inactive substance which does not contain any active ingredients).

ELIGIBILITY:
* At least 2 year history of episodic cluster headache (meeting IHS criteria)
* At least 2 previous episodes
* Expected duration of cluster period is at least 6 weeks but not longer than 24 weeks
* At least 1 but not more than 8 headaches on each of the 3 days immediately prior to treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2003-08; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Phillips, MD, Study Director — Winston Laboratories
Locations (6):
- United States (6):
  - San Francisco Clinical Research Center, San Francisco, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Colorado Neurology and Headache Clinic, Denver, Colorado
  - Diamond Headache Clinic, Chicago, Illinois
  - New York Headache Center, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio